CLINICAL TRIAL: NCT03246022
Title: Huai'an First People's Hospital
Brief Title: Characteristics of Obstructive Sleep Apnea Syndrome Related Hypertension and the Effect of Continuous Positive Airway Pressure Treatment on Blood Pressure
Status: Completed | Type: Observational
Sponsor: Huai'an No.1 People's Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, ZiLi Meng, The director of the of sleep center in Department of Respirology,Huai'an NO.1People's Hospital, Huai'an No.1 People's Hospital
Other Study IDs: Huaian First People's Hospital
Record Dates: First submitted 2017-08-05; First posted 2017-08-11 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-08

CONDITIONS: Hypertension Secondary
Keywords: blood pressure fluctuation; hypertension; continuous positive airway pressure; intermittent hypixa; oxygen desaturation
MeSH Terms: conditions — Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group l: SBP index was less than 30% of AHI
  Interventions: Other: continuous positive airway pressure
- Group 2: SBP index was less than 60% but more than 30%
  Interventions: Other: continuous positive airway pressure

INTERVENTIONS:
Other: continuous positive airway pressure — Continuous positive airway pressure (CPAP) prevents the airway collapse, avoids the occurrence of intermittent hypoxemia and arousal, is the preferred treatment for OSAS and has been widely used in clinical. The investigator would compare the effect of CPAP treatment on awake and sleep BP level at the first night and 2 weeks therapy among three groups. Moreover, whether or not the sympathetic-parasympathetic nerve balance and the renin-angiotensin-aldosterone system are different in three groups would also be evaluated.

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) causes nocturnal chronic intermittent hypoxia (CIH) that contributes to the development of hypertension. CIH profiles, including the its length, speed and intensity were widely different in individuals. Until recently, the influence of OSAS-related IH profiles on hypertension development has not been fully explored. The present study aimed to investigate the effects of different CIH properties on blood pressure (BP) and short-term blood pressure variability (BPV) in severe OSAS patients.

Continuous positive airway pressure (CPAP) prevents the airway collapse, avoids the occurrence of intermittent hypoxemia and arousal, is the preferred treatment for OSAS and has been widely used in clinical. In theory, CPAP maintains upper airway patency and preserves ventilation, thereby inhibits the chain reaction over activation of the sympathetic nervous system and blood pressure regulating mechanism, thus CPAP treatment have adequate scientific basis to cause a substantial reduction arterial blood pressure, but controlled studies showed either no effect or only a minor decrease in arterial blood pressure by 1.4 and 2.5 mmHg respectively.The current, which type of combination of hypertension OSA patients can obtain the best antihypertensive benefit from CPAP therapy is still under debate.

DETAILED DESCRIPTION:
Nocturnal BP was continuously monitored via measurement of pulse transmit time (PTT). The value of apnea-related systolic BP elevation (△BP) was used to reflect short-term BPV. Beat-to-beat RR interval data were incorporated in polysomnography for heart rate variability analysis. LF/HF band ratio was compared between two groups which used to reflect sympatho-vagal balance. The length of the desaturation event was measured to the nearest 0.5 second (△t). The fall in SpO2 during apnea was calculated as the gap from start of the desaturation to the nadir of the desaturation. The rate of fall in SpO2 was counted as the change in the percentage of SpO2 per second (△SpO2 /△t) and expressed as oxygen desaturation rate (ODR), which reflected the speed and efficacy of oxygen desaturation during an apnea event. One hundred and two severe OSAS subjects were divided into two groups according to the their median ODR: faster ODR and slower ODR.

In addtion,patient were categorized into three groups: Group l: systolic blood pressure index was less than 30% of AHI; Group 2: systolic blood pressure index was less than 60% but more than 30%; Group 3: systolic blood pressure index is more than 60% of AHI. The investigator would compare the effect of CPAP treatment on awake and sleep BP level at the first night and 2 weeks therapy among three groups. Moreover, whether or not the sympathetic-parasympathetic nerve balance and the renin-angiotensin-aldosterone system are different in three groups would also be evaluated. The main purpose of study is to confirm the OSA with hypertension and OSA secondary hypertension are two different concepts. Basis for the clinical treatment, the former, CPAP might have no effect or only a minor decrease in arterial blood pressure, while the latter CPAP treatment might achieve significant antihypertensive effect.

ELIGIBILITY:
Inclusion Criteria:

1. BP≤180/110mmHg,but≥140/90mmHg
2. without taking oral antihypertensive drugs. Exclusion criteria.

(1) patients who had been hospitalized for cardiac or respiratory exacerbation<6wk prior to recruiting; (2) with autonomic nervous system diseases or endocrine disorders which might influence BP; (3) unwilling to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. age between 18 to 70 yrs;
  2. newly diagnosed OSAS without treatment;
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
awake systolic blood pressure(SBP)changes | change from Baseline Systolic Blood Pressure at 2 weeks
  as the mean systolic blood pressure measurements during a supine resting period of 1 0minute at awake state
sleep systolic blood pressure(SBP)changes | change from Baseline Systolic Blood Pressure at 2 weeks
  as the average of systolic blood pressure values during sleep
sympathetic-parasympathetic nerve balance changes | change from Baseline Systolic Blood Pressure at 2 weeks
  Studies using spectral analysis of R-R intervals have reported that the power spectrum contains both low-frequency(LF,0.04-0.15 Hz)and high-frequency peaks(HF,0.15-0.5Hz),HF power reflects parasympathetic activity,whereas LF power primarily reflects sympathetic activity with a parasympathetic component.The LF-to-HF ratio(LF/HF)is commonly regarded as an index of sympathovagal balance
renin-angiotensin-aldosterone systemchanges | change from Baseline Systolic Blood Pressure at 2 weeks
  as the levels of plasma angiotension ⅰ( Ang I) and angiotension ⅱ( Ang ⅱ) before and after CPAP treatment
AHI changes | change from Baseline Systolic Blood Pressure at 2 weeks
  the combined number of apnea and hypopnea episodes per hour of sleep
TST90 changes | change from Baseline Systolic Blood Pressure at 2 weeks
  percentage of sleep time with oxygen saturation < 90%
oxygen desaturation index（ODI） changes | change from Baseline Systolic Blood Pressure at 2 weeks
  oxygen desaturation index
event-related systolic blood pressure elevation (△SBP) changes | change from Baseline Systolic Blood Pressure at 2 weeks
  as the gap between the peak value of postapneic SBP and lowest SBP during a obstructive respiratory event
systolic blood pressure(SBP)index | change from Baseline Systolic Blood Pressure at 2 weeks
  as the number of △SBP>10mmHg per hour of sleep time.
Desaturation rate | one night
  The rate of fall in SpO2 was counted as the change in the percentage of SpO2 per second during apnea

CONTACTS AND LOCATIONS:
Overall Officials: Zili Meng, Master, Study Director — Department Of Respiratory Medicine,Huai'an First People's Hospital,Nanjing Medical University
Locations (1):
- Department Of Respiratory Medicine,Huai'an First People's Hospital,Nanjing Medical University, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meng Z, Chen Y, Yang T, Sun B, Luo C, Wei G, Xie X, Gu Y, Ding N, Zhang X, Xu J. New perspective on exploring the predictive factors of blood pressure reduction during CPAP treatment in people with severe OSA and hypertension: a prospective observational study. BMJ Open Respir Res. 2023 May;10(1):e001560. doi: 10.1136/bmjresp-2022-001560. PMID 37169401
- [Derived] Wang N, Meng Z, Ding N, Chen W, Zhang X, Huang M, Xu J. Oxygen desaturation rate as a novel intermittent hypoxemia parameter in severe obstructive sleep apnea is strongly associated with hypertension. J Clin Sleep Med. 2020 Jul 15;16(7):1055-1062. doi: 10.5664/jcsm.8396. PMID 32105212